CLINICAL TRIAL: NCT00201370
Title: A Multi-center Survey of HPV in Cervical Intraepithelial Neoplasia (CIN) With Longitudinal Follow-up of LSIL Cases
Status: Completed | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: T1899
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2005-09

CONDITIONS: Cervical Cancer; Low-grade Squamous Intraepithelial Lesion,; Human Papillomavirus
Keywords: cervical neoplasia;; human papillomavirus,; PCR,; risk factors,; Taiwan
MeSH Terms: conditions — Uterine Cervical Neoplasms; Squamous Intraepithelial Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aims of this study are:

1. Surveillance of the prevalence of HPV infection in ASCUS, AGCUS and SIL cases pooled from medical centers in Taiwan and analysis of the related epidemiological factors.
2. Providing a better understanding of the natural history of HPV infection with its correlation with pathologic changes through a longitudinal follow-up of LSIL cases.

DETAILED DESCRIPTION:
Carcinoma of the uterine cervix is by far the most prevalent cancer of women in Taiwan and worldwide. In 1994, it ranked the top of female cancer incidence with 3000 new cases annually and claimed nearly 1000 lives. The major cause of this malignant disease is now pointed to the infection of oncogenic types of human papillomavirus (HPV). HPV infection is sexually transmitted, affects the immature metaplastic cells of uterine cervix and, in an unknown proportion, results in squamous intraepithelial lesion (SIL) of differing severity. The natural history of HPV infection is by far elusive. It is not clear how the virus get into the cell, how the immune system respond to it, and how the epithelial cell get transformed. An average estimation holds that about 60% of low grade SIL will regress, 30% will persist, 10% will progress to high grade lesions and less than 1% become invasive lesions.

The aims of this study are:

1. Surveillance of the prevalence of HPV infection in ASCUS, AGCUS and SIL cases pooled from medical centers in Taiwan and analysis of the related epidemiological factors.
2. Providing a better understanding of the natural history of HPV infection with its correlation with pathologic changes through a longitudinal follow-up of LSIL cases.

Through a consensus of management of patients with abnormal Pap smear in TGOG, a standard protocol of specimen collection, clinical follow-up has been established. Patients with a Pap smear of ASCUS, AGCUS or SIL will be arranged with a repeat Pap smear and a colposcopy with or without biopsy. A cervical swab will be taken and sent to the core laboratory for HPV DNA detection and genotyping. Pap smear and biopsies were then panel-reviewed by Pathologists. Cytology-or pathology-proved LSIL cases will be followed every three months with Pap smear, colposcopy and HPV test until disease progression or two consecutive negative results of all the three data. One thousand cases fulfilling "aim 1" will be analyzed during the first year, and the nature course of about 300 LSIL cases will be followed at the end of the third year.

ELIGIBILITY:
Inclusion Criteria:

* Women visiting the gynecologic clinic of the participating medical centers and have a recent (within three months) Pap smear result of ASCUS, AGCUS, LSIL and HSIL of during the study period will be invited to this study.
* An informed consent signed.

Exclusion Criteria:

- Women who are not pregnant, had had no previous CIN

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women were invited to participate in the cross-sectional study
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 1999-08; Primary Completion 2004-02 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the disease-free survival. | 5

SECONDARY OUTCOMES:
Secondary endpoints include overall survival and tumor response rate. | 5

CONTACTS AND LOCATIONS:
Overall Officials: Tang-Yuan Chu, M.D., Ph.D., Principal Investigator — Taiwan cooperative oncology group
Locations (4):
- Taiwan (4):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Tri-Services General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Chang-Gung Memorial Hospital(Lin-Kou),, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Journal of Medical Virology Volume 77, Issue 2, pages 273-281, October 2005
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/16121376?ordinalpos=20&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum